CLINICAL TRIAL: NCT03486691
Title: Preoperative Ultrasonographic Liver Size as a Predictor for Difficulty in Bariatric Surgery
Brief Title: Preoperative Ultrasound as a Predictor for Difficulty in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fac.med.055
Record Dates: First submitted 2018-03-07; First posted 2018-04-03 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative left lobe measurement (Experimental): routine preoperative left lobe measurement
  Interventions: Other: Routine measurement of left lobe
- Control group (Active Comparator): Control group without routine measurement of left lobe
  Interventions: Other: control group

INTERVENTIONS:
Other: Routine measurement of left lobe — Routine preoperative measurement of left lobe
  Arms: preoperative left lobe measurement
Other: control group — no routine preoperative measurement of left lobe
  Arms: Control group

SUMMARY:
the left lobe of the liver in obese patient usually fatty and enlarged and may cause difficulty during bariatric surgery. the aim of this study is to test the impact of routine preoperative ultrasound to evaluate the size of left lobe of the liver as a preoperative predictor for difficulty

DETAILED DESCRIPTION:
the left lobe of the liver in obese patient usually fatty and enlarged and may cause difficulty during bariatric surgery. the aim of this study is to test the impact of routine preoperative ultrasound to evaluate the size of left lobe of the liver as a preoperative predictor for difficulty. two equal groups of patients are operated by laparoscopic sleeve gastrectomy with loop bipartition, in one group routine abdominal ultrasound is done, in the other group ultrasound not routinely done.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patient with BMI more than 40 with or without co-morbidity
* Morbidly obese patient with BMI more than 35 with co-morbidity

Exclusion Criteria:

* Unfit patients for laparoscopy
* patients refuse to share in the study
* revisional surgery for obesity
* previous upper abdominal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
intraoperative maximum diameter of left lobe of the liver | 4 hours
  intraoperative maximum diameter of left lobe of the liver in centimeter using intraoperative tape
score of difficulty | 6 hours
  score of difficulty from:exposure of the hiatus, retraction of the liver and operative time

SECONDARY OUTCOMES:
operative time | 6 hours
  operative time from skin to skin
incidence of intraoperative complications | 3 days
  incidence of intraoperative complications like bleeding,or injury to intra-abdominal organ
early postoperative complications | 2 weeks
  early postoperative complications like leak or vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Sewefy, Principal Investigator — Minia University
Locations (1):
- Faculty of medicine, Minya, Egypt